CLINICAL TRIAL: NCT01860963
Title: Prevalence of Anal Dysplasia in Patients With Inflammatory Bowel Disease and Healthy Controls
Brief Title: Anal Dysplasia in Patients With Inflammatory Bowel Disease and Healthy Controls
Acronym: ADIBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: MW-16467
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Anal Squamous Intraepithelial Lesion (ASIL); HPV DNA
Keywords: ASIL; Anal dysplasia; IBD; HPV DNA

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- IBD patients on immunosuppression (Active Comparator): Patients on azathioprine/6-mercaptopurine (6MP), prednisone, methotrexate, infliximab, adalimumab, certolizumab, natalizumab, and etanercept are included.
  Interventions: Procedure: Anal Pap smear and HPV DNA testing
- IBD patients off immunosuppressants (Active Comparator): Patients off immunosuppressants, on 5-aminosalicylic acid (5-ASA) agents, antibiotics, or no treatment for IBD are included.
  Interventions: Procedure: Anal Pap smear and HPV DNA testing
- Healthy controls (Active Comparator): Age-matched healthy controls enrolled from the hospital, outpatient clinics, and from the general public via flyers and online advertisements.
  Interventions: Procedure: Anal Pap smear and HPV DNA testing

INTERVENTIONS:
Procedure: Anal Pap smear and HPV DNA testing — Anal Pap smear is a standard diagnostic test used for early detection of pre-cancerous cells and anal HPV.

SUMMARY:
This study is designed to establish the prevalence of anal squamous intraepithelial lesion (ASIL) in patients with inflammatory bowel disease (IBD) and healthy controls.

DETAILED DESCRIPTION:
IBD patients attending the Stanford Inflammatory Bowel Disease (IBD) clinic and age-matched healthy controls are screened for eligibility. Informed consent is obtained for eligible subjects. An anonymous self-administered questionnaire is administered to assess risk factors for HPV. For IBD patients, information regarding IBD diagnosis and treatment is obtained.

An anal pap smear is performed at the time of a clinic visit or at the time of an already scheduled colonoscopy. Samples are collected and processed at Stanford pathology where a blinded pathologist reads all specimens. Human Papillomavirus (HPV) DNA testing is performed on all specimens. All patients with anal squamous intraepithelial lesion (ASIL) are referred to a colorectal surgeon for further recommendations or treatment, which includes a high-resolution anoscopy.

ELIGIBILITY:
Inclusion Criteria:

* All IBD patients followed in the IBD clinic and healthy controls who are greater than 18 years old

Exclusion Criteria:

* History of HPV vaccination
* Pregnancy
* Other immunosuppressed states (i.e. systemic lupus erythematosus, rheumatoid arthritis, cancer, Human Immunodeficiency Virus (HIV), transplant)
* IBD patients who don't meet immunosuppression/non-immunosuppression criteria
* Inability to obtain informed consent from patient
* Previous diagnosis of ASIL or anal/rectal cancer

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Presence of high risk HPV and/or abnormal cytology | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Mark Welton, MD, Principal Investigator — Stanford Hosptial and Clinics; Shamita Shah, MD, Principal Investigator — Stanford Hospital and Clinics
Locations (1):
- Stanford Digestive Health Center, Stanford, California, United States

REFERENCES:
- [Derived] Shah SB, Pickham D, Araya H, Kamal A, Pineda CE, Ghole S, Shih L, Kong C, Pai R, Welton M. Prevalence of Anal Dysplasia in Patients With Inflammatory Bowel Disease. Clin Gastroenterol Hepatol. 2015 Nov;13(11):1955-61.e1. doi: 10.1016/j.cgh.2015.05.031. Epub 2015 Jun 2. PMID 26044314